CLINICAL TRIAL: NCT01563744
Title: EGD-assisted Bowel Preparation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockford Gastroenterology Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGD-assisted 2012
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Esophagoscopy Techniques; Colonoscopy
Keywords: colonoscopy; bowel preparation; tolerability; EGD-assisted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGD-assisted colonoscopy prep (Experimental): 2 liters of polyethylene glycol instilled through the channel of the endoscope during EGD when colonoscopy expected the following day. Patients follow a clear liquid diet, then ingest an addition 1 liter polyethylene glycol 4 hours prior to colonoscopy. Patients are also given a tap water enema 1 hour prior to colonoscopy.
  Interventions: Procedure: EGD-assisted administration of colonoscopy prep
- Standard Colonoscopy Prep (Active Comparator): Split-dose polyethylene glycol (2 liters pm prior to colonoscopy, 1 liter 4 hours prior to colonoscopy)), clear liquid diet, metoclopramide 10 mg IV 30 minutes prior to procedure, tap water enema 1 hr prior to colonoscopy
  Interventions: Procedure: Control Group received standard prep by oral administration

INTERVENTIONS:
Procedure: EGD-assisted administration of colonoscopy prep — Interventional group receive the first 2 liters of prep solution during EGD through the scope channel if colonoscopy expected the following day.
  Arms: EGD-assisted colonoscopy prep
Procedure: Control Group received standard prep by oral administration — Control group receive standard oral colonoscopy prep.
  Arms: Standard Colonoscopy Prep

SUMMARY:
Adequate bowel preparation is of critical importance for colonoscopy. Particularly among hospitalized patients, inadequate bowel preparation for colonoscopy may arise due to patient intolerance to prescribed laxative regimen, elderly population, and co-existing conditions that impair the ability to ingest a large-volume laxative regimen. Improvements in bowel preparation for colonoscopy in hospitalized patients would likely improve patient care and reduce hospital costs. The purpose of this study is to determine if administering a portion of the bowel purgative via EGD could improve colonoscopy preparation in hospitalized patients.

DETAILED DESCRIPTION:
In this randomized controlled trial in hospitalized patients, patients in whom colonoscopy was anticipated the day following EGD were consented and randomized to either standard prep by mouth (split-dose PEG) or intervention group (instillation of the first 2 liters of Nulytely solution through the channel of the endoscope into the duodenal bulb, then continue standard prep). Data is collected on quality of prep and patient satisfaction in both groups.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients
* having EGD and expected to have colonoscopy the following day
* written informed consent

Exclusion Criteria:

* unable to tolerate EGD-assisted prep administration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | Twenty four to 48 hours - from time of consent prior to EGD until end of colonoscopy performed the following day
  Quality of prep was assessed using the Ottawa bowel preparation scale (Rostom A, Jolicoeur E. Validation of a new scale for the assessment of bowel preparation quality. Gastrointest endosc 2004;59:482-6)

SECONDARY OUTCOMES:
Patient tolerance of bowel preparation | administered just prior to sedation for colonoscopy
  Patients in both groups were asked to indicate if the bowel prep was easy, slightly difficult, moderately difficult, extremely difficult, or if they were unable to complete the prep as directed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Barclay, MD, Principal Investigator — Rockford Gastroenterology Associates, University of Illinois College of Medicine, Rockford
Locations (2):
- United States (2):
  - SwedishAmerican Hospital, Rockford, Illinois
  - St. Anthony Medical Center, Rockford, Illinois

IPD SHARING:
Plan to Share IPD: No